CLINICAL TRIAL: NCT07123857
Title: Impact of Point-of-care Lactate Testing as Triage Supplement on Patient Management Using Manchester Triage System
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University Medical Centre Maribor (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Screening
Other Study IDs: IRP-2024/01-13
Record Dates: First submitted 2025-07-16; First posted 2025-08-14 (Actual); Last update posted 2025-08-14 (Actual); Status verified 2025-08

CONDITIONS: Triage; Emergency Department Triage; Emergency Department Overcrowding; Emergency Medicine

STUDY DESIGN:
Who Masked: Participant, Care Provider
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Control group - No-retriage (No Intervention)
- Test group - Retriage to orange MTS group (Experimental)
  Interventions: Diagnostic Test: re-triage

INTERVENTIONS:
Diagnostic Test: re-triage — Patients in the test group will be re-triaged into the orange MTS category.
  Arms: Test group - Retriage to orange MTS group

SUMMARY:
Although the Manchester Triage System (MTS) is widely used and validated internationally, it has some limitations. Its accuracy is moderate, especially for children and the elderly. Rising patient numbers and overcrowded emergency departments increase wait times, sometimes beyond safe limits. In Slovenia, MTS has been in use for 14 years without major updates, despite a significant rise in emergency visits. The yellow triage category (60-minute wait time) includes a very diverse group of patients, some of whom might require faster care. Older patients, in particular, often show atypical symptoms and may be under-triaged. Including rapid bedside lab tests, like blood lactate levels, could improve risk assessment and triage accuracy. Elevated lactate is linked with higher mortality and can help identify critically ill patients more effectively. The proposed study is a prospective, randomized trial involving two groups of patients in the yellow triage category, all of whom will have their capillary blood lactate levels measured. Patients with normal lactate levels will be excluded. Only patients with elevated lactate will be compared. The test group will be re-triaged to the orange category and treated more urgently. The control group, despite also having high lactate levels, will remain in the yellow category, and their elevated lactate values will not be shared with the treating physician. Randomization will be based on the patient's birth date (even days = test group, odd days = control group). Only the nurse will know the result, maintaining physician blinding to avoid the Hawthorne effect-changes in behavior due to awareness of being studied. Standard lab tests will be performed later during treatment as deemed necessary by the attending doctor.

ELIGIBILITY:
Inclusion Criteria:

* signed consent, yellow MTS triage category

Exclusion Criteria:

* pregnant women, trauma patients, epileptic seizures, adrenergic therapy in prehospital unit

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 200 (Estimated)
Dates: Start 2025-07-10 (Actual); Primary Completion 2026-12-31 (Estimated); Study Completion 2026-12-31 (Estimated)

PRIMARY OUTCOMES:
Vasoactive drug use | 30-day

SECONDARY OUTCOMES:
In-hospital mortality | 30-day
ICU admission | 30-day

CONTACTS AND LOCATIONS:
Locations (1):
- University Medical Center Maribor, Maribor, Slovenia

IPD SHARING:
Plan to Share IPD: No
Individual participant data will not be shared with other researchers. The decision not to share IPD is based on privacy concerns, data protection regulations, and institutional policy.